CLINICAL TRIAL: NCT00199524
Title: A Prospective Randomized Controlled Clinical Trial of the Use of a Ureteral Access Sheath During Ureteroscopy and Its Effect on Stone Free Rate
Brief Title: Use of a Ureteral Access Sheath During Ureteroscopy and Its Effect on Stone Free Rate
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was slower than anticipated.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Dr. Hassan Razvi, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-05-002
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Urinary Calculi
Keywords: ureteroscopy; stone free
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ureteroscopy with ureteral access sheath
  Interventions: Device: Navigator Ureteral Access Sheath
- 2 (No Intervention): ureteroscopy without ureteral access sheath

INTERVENTIONS:
Device: Navigator Ureteral Access Sheath — ureteral access sheath
  Other Names: Navigator Ureteral Access Shealth
  Arms: 1

SUMMARY:
Patients with upper ureteral or renal stones will be randomized to undergoing ureteroscopy with or without a ureteral access sheath. The sheath is designed to facilitate ureteroscope insertion and re-insertion, thus allowing fragments to be basketed out. Stone free rates at 3 months will be determined between the two groups.

The investigators hypothesize that the use of the ureteral access sheath with ureteroscopy will result in improved stone free rates at 3 months compared to ureteroscopy without use of a sheath.

ELIGIBILITY:
Inclusion Criteria:

* Upper ureteral (proximal to iliac vessels/iliac crest) calculi;
* Renal calculi;
* Normal renal function;
* Any stone composition;
* Single or multiple stones(planned treatment of all stones at this surgery);
* Age > 18 years;
* Able and willing to return treatment centre for follow-up visits; AND
* Signed study consent

Exclusion Criteria:

* Ureteric calculi distal to the level of the iliac vessels/iliac crest;
* Failed ureteroscopy for same stone (i.e. has to be the first ureteroscopic procedure for this stone, however a prior failed extracorporeal shockwave lithotripsy (SWL) is acceptable);
* Bilateral ureteroscopy;
* If an adjunctive procedure is planned post ureteroscopy (e.g. percutaneous nephrolithotomy, SWL) (i.e. it is known preoperatively that a ureteroscopic procedure will not render the patient stone free and that ancillary procedures will be necessary);
* If in the investigators opinion, enrollment would be not be appropriate; OR
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary end point is the stone free rate at 3 months post ureteroscopy. | 3 months post ureteroscopy

SECONDARY OUTCOMES:
Secondary end points include operative and surgical factors such as operative time, stone size, stone location, stone composition, patient sex and the presence of a ureteric stent post-op. | at time of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Razvi, MD, FRCSC, Principal Investigator — Urology, St. Joseph's Hospital, The University of Western Ontario
Locations (5):
- Canada (5):
  - Edmonton Prostate and Urological Research Centre, Edmonton, Alberta
  - The Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - Centre for Advanced Urological Research at Queen's University, Kingston, Ontario
  - Urology at St. Joseph's Hospital, The University of Western Ontario, London, Ontario
  - Kidney Stone Program at St. Michael's Hospital, Toronto, Ontario